CLINICAL TRIAL: NCT01685203
Title: A Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Coadministration of ABT-450 With Ritonavir (ABT-450/r) and ABT-267 in Adults With Chronic Hepatitis C Virus Infection (PEARL-I)
Brief Title: A Study to Evaluate the Safety and Effect of Co-administration of ABT-450 With Ritonavir (ABT-450/r) and ABT-267 in Adults With Chronic Hepatitis C Virus Infection
Acronym: PEARL-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-393; 2011-005762-38 (EudraCT Number)
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C Virus; Ribavirin-Free; Hepatitis C Genotype 1; Hepatitis C; Interferon-Free; Chronic Hepatitis C; Compensated cirrhosis; Hepatitis C Genotype 4; Paritaprevir; Ombitasvir; Ritonavir; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — paritaprevir; ombitasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1 (Experimental): ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 12 weeks to adult noncirrhotic, treatment-naïve, HCV GT4-infected participants
  Interventions: Drug: ABT-450/r; Drug: ABT-267
- Group 2 (Experimental): ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 12 weeks to adult noncirrhotic, treatment-naïve HCV GT1b-infected participants
  Interventions: Drug: ABT-450/r; Drug: ABT-267
- Group 3 (Experimental): ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 12 weeks to adult noncirrhotic, HCV GT1b-infected, pegylated-interferon/ribavirin (pegIFN/RBV) treatment null responder participants
  Interventions: Drug: ABT-450/r; Drug: ABT-267
- Group 4 (Experimental): ABT-450 150 mg/ r 100 mg, ABT-267 25 mg , once daily and weight-based ribavirin (RBV; 1,000 mg/day if < 75 kg or 1,200 mg/day if ≥ 75 kg, divided twice daily) for 12 weeks to adult noncirrhotic, treatment-naïve, HCV GT4-infected participants
  Interventions: Drug: ABT-450/r; Drug: ABT-267; Drug: Ribavirin (RBV)
- Group 5 (Experimental): ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 12 weeks to adult noncirrhotic, treatment-experienced, HCV GT4-infected participants
  Interventions: Drug: ABT-450/r; Drug: ABT-267
- Group 6 (Experimental): ABT-450 150 mg/ r 100 mg, ABT-267 25 mg , once daily and weight-based ribavirin (RBV; 1,000 mg/day if < 75 kg or 1,200 mg/day if ≥ 75 kg, divided twice daily) for 12 weeks to adult noncirrhotic, HCV GT4-infected, pegylated-interferon/RBV (pegIFN/RBV) treatment-experienced participants
  Interventions: Drug: ABT-450/r; Drug: ABT-267; Drug: Ribavirin (RBV)
- Group 7 (Experimental): ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 24 weeks to adult, HCV GT1b-infected, treatment-naïve participants with compensated cirrhosis
  Interventions: Drug: ABT-450/r; Drug: ABT-267
- Group 8 (Experimental): ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 24 weeks to adult, HCV GT1b-infected, pegylated-interferon/RBV(pegIFN/RBV) treatment-experienced participants with compensated cirrhosis
  Interventions: Drug: ABT-450/r; Drug: ABT-267

INTERVENTIONS:
Drug: ABT-450/r — Tablet; ABT-450; Capsule; ritonavir
  Other Names: ABT-450 also known as paritaprevir
Drug: ABT-267 — Tablet
  Other Names: ABT-267 also known as ombitasvir
Drug: Ribavirin (RBV) — Tablet
  Arms: Group 4; Group 6

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of co-administration of ABT-450 (also known as paritaprevir) with ritonavir (ABT-450/r) and ABT-267 (also known as ombitasvir) in adults with chronic hepatitis C virus infection.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, open-label, combination treatment study of the 2-DAA regimen (ABT-450 150 mg QD + ritonavir 100 mg QD + ABT-267 25 mg QD) in adult HCV GT1b-infected treatment-naïve and Pegylated-interferon/ribavirin (pegIFN/RBV) treatment-experienced participants without cirrhosis and with compensated cirrhosis, and in adult GT4-infected treatment-naïve and pegIFN/RBV treatment-experienced participants without cirrhosis. Treatment Group 5 was not open to enrollment, based on a protocol-specified interim review of results from the treatment-naïve GT4 Groups 1 and 4 that indicated higher sustained virologic response (SVR) rates among participants receiving the 2-DAA regimen with RBV. All other groups completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be postmenopausal for more than 2 years or surgically sterile
* Subjects must meet one of the following:

  * Treatment-naive: Subject has never received antiviral treatment for hepatitis C infection OR
  * Treatment Experienced (Prior null responders, Partial responders or Relapsers to pegIFN/RBV);
* Body mass index (BMI) is ≥ 18 to < 38 kg/m^2.
* Chronic HCV genotype 1b infection/with or without cirrhosis or HCV genotype 4 infection/without cirrhosis for at least 6 months prior to study screening.
* Subject has plasma HCV RNA level > 10,000 IU/mL at Screening

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any drug.
* Females who were pregnant or planned to become pregnant, or breastfeeding, or GT4-infected males whose partners were pregnant or planning to become pregnant within 7 months (or per local RBV label) after their last dose of study drug/RBV.
* Recent history of drug or alcohol abuse that could preclude adherence to the protocol.
* Positive test result for hepatitis B surface antigen or anti-Human Immunodeficiency Virus (HIV) antibodies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilou Mobashery, MD, Study Director — AbbVie

REFERENCES:
- [Background] Hezode C, Asselah T, Reddy KR, Hassanein T, Berenguer M, Fleischer-Stepniewska K, Marcellin P, Hall C, Schnell G, Pilot-Matias T, Mobashery N, Redman R, Vilchez RA, Pol S. Ombitasvir plus paritaprevir plus ritonavir with or without ribavirin in treatment-naive and treatment-experienced patients with genotype 4 chronic hepatitis C virus infection (PEARL-I): a randomised, open-label trial. Lancet. 2015 Jun 20;385(9986):2502-9. doi: 10.1016/S0140-6736(15)60159-3. Epub 2015 Mar 31. PMID 25837829
- [Background] Lawitz E, Makara M, Akarca US, Thuluvath PJ, Preotescu LL, Varunok P, Morillas RM, Hall C, Mobashery N, Redman R, Pilot-Matias T, Vilchez RA, Hezode C. Efficacy and Safety of Ombitasvir, Paritaprevir, and Ritonavir in an Open-Label Study of Patients With Genotype 1b Chronic Hepatitis C Virus Infection With and Without Cirrhosis. Gastroenterology. 2015 Oct;149(4):971-80.e1. doi: 10.1053/j.gastro.2015.07.001. Epub 2015 Jul 11. PMID 26170136
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study originally planned to enroll Group 5 (GT4 treatment-experienced, 2-DAA regimen for 12 weeks), but based on a protocol-specified interim review of results from the treatment-naïve GT4 Groups 1 and 4 that indicated higher SVR rates among participants receiving the 2-DAA regimen with RBV, Group 5 was not opened to enrollment.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Started | 44 | 42 | 40 | 42 | 49 | 47 | 52
Completed Study Drug | 42 | 40 | 39 | 42 | 49 | 43 | 52
Completed | 40 | 39 | 40 | 41 | 49 | 44 | 52
Not Completed | 4 | 3 | 0 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse event and withdrew consent | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient's decision | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8 | Total
Number analyzed (Participants) | 44 | 42 | 40 | 42 | 49 | 47 | 52 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (10.0) | 55.8 (6.9) | 54.2 (9.6) | 44.2 (12.7) | 50.9 (10.1) | 57.8 (7.1) | 57.1 (6.0) | 52.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 25 | 14 | 13 | 24 | 19 | 132
  Male | 24 | 25 | 15 | 28 | 36 | 23 | 33 | 184

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants in Each Treatment Group With Sustained Virologic Response 24 Weeks Post-treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [<LLOQ]) 24 weeks after the last dose of study drug.
Time Frame: 24 weeks after the last actual dose of study drug
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 44 | 42 | 40 | 42 | 49 | 47 | 52
Percentage of participants | 86.4 [72.6 to 94.8] | 92.9 [80.5 to 98.5] | 90.0 [76.3 to 97.2] | 100.0 [91.6 to 100.0] | 100.0 [92.7 to 100.0] | 97.9 [88.7 to 99.9] | 98.1 [89.7 to 100.0]

2. Primary Outcome: Percentage of Participants in Each Treatment Group With Sustained Virologic Response 12 Weeks Post-treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 44 | 42 | 40 | 42 | 49 | 47 | 52
Percentage of participants | 90.9 [78.3 to 97.5] | 95.2 [83.8 to 99.4] | 90.0 [76.3 to 97.2] | 100 [91.6 to 100.0] | 100 [92.7 to 100.0] | 97.9 [88.7 to 99.9] | 98.1 [89.7 to 100.0]
Statistical Analysis 1: Comparison: Group 2 vs Group 3; Test type: Superiority or Other; p = 0.381, Regression, Logistic; Treatment group, baseline log(subscript)10(subscript) HCV RNA level and Interleukin-28B (IL28B) genotype (CC or non-CC) were used as predictors
Statistical Analysis 2: Comparison: Group 1 vs Group 4; Test type: Superiority or Other; p = 0.086, Stratum-adjusted Mantel-Haenszel — Difference in rates after adjusting for Interleukin-28 (IL28) genotype (CC or Non-CC) using stratum-adjusted Mantel-Haenszel proportions and continuity-corrected variances

3. Secondary Outcome: Percentage of Participants in Each Treatment Group With On-treatment Virologic Failure.
Description: Virologic failure during treatment was defined as rebound (confirmed HCV RNA greater than or equal to the lower limit of quantitation [≥ LLOQ] after HCV RNA < LLOQ during treatment, or confirmed increase from the lowest value post baseline in HCV RNA [2 consecutive HCV RNA measurements > 1 log(subscript)10(subscript) IU/mL above the lowest value post baseline] at any time point during treatment), or fail to suppress (HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks [≥ 36 days] of treatment).
Time Frame: Baseline (Day 1), Day 3, and Treatment Weeks 1, 2 ,3 ,4, 6, 8, 10, and 12 for all participants and Treatment Weeks 16, 20 and 24 for Groups 7 and 8
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 44 | 42 | 40 | 42 | 49 | 47 | 52
Percentage of participants | 2.3 [0.1 to 12.0] | 0 [0.0 to 8.4] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.4] | 0 [0.0 to 7.3] | 0 [0.0 to 7.5] | 0 [0.0 to 6.8]

4. Secondary Outcome: Percentage of Participants in Each Treatment Group With Post-treatment Virologic Relapse.
Description: Participants were considered to have virologic relapse after treatment if they had confirmed quantifiable plasma Hepatitis C virus ribonucleic acid (HCV RNA) ≥ lower limit of quantification (LLOQ) between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA < LLOQ at the end of treatment.
Time Frame: Within 12 weeks after the last dose of study drug
Population: All randomized participants who received at least 1 dose of study drug and completed treatment with HCV RNA < LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 42 | 40 | 39 | 42 | 49 | 44 | 52
Percentage of participants | 4.8 [0.6 to 16.2] | 0 [0.0 to 8.8] | 7.7 [1.6 to 20.9] | 0 [0.0 to 8.4] | 0 [0.0 to 7.3] | 0 [0.0 to 8.0] | 1.9 [0.0 to 10.3]

5. Secondary Outcome: Percentage of Participants in Each Treatment Group With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events were defined as any event that began or worsened in severity after initiation of study drug through 30 days after the last dose of study drug.
Time Frame: From the start of study drug administration until 30 days after the last dose,16 weeks for Groups 1, 2, 3, 4, and 6, and 28 weeks for Groups 7 and 8.
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 44 | 42 | 40 | 42 | 49 | 47 | 52
Percentage of participants | 77.3 | 73.8 | 80.0 | 88.1 | 85.7 | 85.1 | 71.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 30 days after the last dose, 16 weeks for Groups 1, 2, 3, 4, and 6, and 28 weeks for Groups 7 and 8.
Description: Serious adverse events were collected from the time of informed consent until the end of participation, up to 65 weeks.
Groups:
- Group 6: ABT-450 150 mg/ r 100 mg, ABT-267 25 mg , once daily and weight-based ribavirin (RBV; 1,000 mg/day if < 75 kg or 1,200 mg/day if 75 kg, divided twice daily) for 12 weeks to adult noncirrhotic, HCV GT4-infected, pegylated-interferon/ RBV (pegIFN/RBV) treatment-experienced participants
- Group 8: ABT-450 150 mg/ r 100 mg, and ABT-267 25 mg once daily for 24 weeks to adult, HCV GT1b-infected, pegylated-interferon/ RBV(pegIFN/RBV) treatment-experienced participants with compensated cirrhosis
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 6 | Group 7 | Group 8
Serious Adverse Events (participants affected / at risk) | 2/44 | 1/42 | 1/40 | 0/42 | 0/49 | 3/47 | 2/52
Other Adverse Events (participants affected / at risk) | 30/44 | 24/42 | 26/40 | 32/42 | 38/49 | 34/47 | 33/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=44) | Group 2 (N=42) | Group 3 (N=40) | Group 4 (N=42) | Group 6 (N=49) | Group 7 (N=47) | Group 8 (N=52)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEVICE EXTRUSION (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=44) | Group 2 (N=42) | Group 3 (N=40) | Group 4 (N=42) | Group 6 (N=49) | Group 7 (N=47) | Group 8 (N=52)
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 3 | 1 | 0 | 0 | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 3 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 4
DIARRHOEA (Gastrointestinal disorders) | 2 | 6 | 0 | 6 | 3 | 7 | 7
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 4 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3
NAUSEA (Gastrointestinal disorders) | 4 | 8 | 0 | 7 | 6 | 5 | 5
VOMITING (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 0 | 2 | 1
ASTHENIA (General disorders) | 11 | 3 | 2 | 10 | 16 | 10 | 7
FATIGUE (General disorders) | 3 | 6 | 0 | 5 | 9 | 4 | 6
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 2
IRRITABILITY (General disorders) | 3 | 0 | 0 | 6 | 2 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 3 | 0 | 1 | 2 | 2 | 2
PYREXIA (General disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 3 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 1 | 2
NASOPHARYNGITIS (Infections and infestations) | 2 | 1 | 2 | 2 | 6 | 4 | 4
RHINITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 2 | 1 | 2 | 4
URINARY TRACT INFECTION (Infections and infestations) | 3 | 2 | 2 | 1 | 2 | 2 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 3 | 2 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1 | 4 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 4 | 6 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 5 | 3 | 2
DIZZINESS (Nervous system disorders) | 1 | 1 | 3 | 0 | 3 | 0 | 1
HEADACHE (Nervous system disorders) | 13 | 14 | 10 | 14 | 14 | 9 | 10
ANXIETY (Psychiatric disorders) | 2 | 0 | 0 | 4 | 2 | 1 | 2
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 1
INSOMNIA (Psychiatric disorders) | 2 | 1 | 0 | 4 | 8 | 3 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2 | 4 | 3 | 5
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 3
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 7 | 0 | 0 | 3 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 6 | 0 | 1 | 5 | 8 | 9
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.